CLINICAL TRIAL: NCT06576245
Title: Efficacy of Quantum Molecular Resonance Combined With Intense Pulsed Light in Mixed Dry Eye: A Prospective Clinical Study.
Brief Title: Efficacy of Quantum Molecular Resonance Combined With Intense Pulsed Light in Mixed Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, José-María Sánchez-González, Head of Vision Science Research Group, University of Seville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USeville_2024_01
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye
Keywords: Mixed Dry Eye; Quantum Molecular Resonance (QMR); Intense Pulsed Light (IPL); Tear Film Stability; Dry Eye Treatment
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Therapeutics; Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Treatment: Quantum Molecular Resonance (QMR) and Intense Pulsed Light (IPL) (Experimental): Participants in this arm will receive a combination treatment consisting of Quantum Molecular Resonance (QMR) therapy and Intense Pulsed Light (IPL) therapy. The treatment protocol includes 4 sessions of QMR and 3 sessions of IPL over a period of 6 weeks. QMR and IPL will be combined in certain weeks, with additional sessions of QMR and IPL performed separately in other weeks. The effectiveness of this combination therapy will be evaluated through various clinical endpoints, including improvements in tear film stability and dry eye symptoms over a 3-month follow-up period.
  Interventions: Device: Quantum Molecular Resonance (QMR) Therapy; Device: Intense Pulsed Light (IPL) Therapy; Drug: Tear Substitute Treatment (Supportive Therapy)

INTERVENTIONS:
Device: Quantum Molecular Resonance (QMR) Therapy — Quantum Molecular Resonance (QMR) therapy will be administered using the RexonEye® device (Resono Ophthalmic, Trieste, Italy). The device delivers low-intensity, high-frequency electrical waves ranging from 4-64 MHz through specialized contact electrodes. Participants will receive 4 QMR treatment sessions over 6 weeks. Each session lasts for 20 minutes, with a 30-second alternation between the eyes. The goal of QMR therapy is to stimulate cellular regeneration and improve tear production by targeting the lacrimal gland.
Device: Intense Pulsed Light (IPL) Therapy — Intense Pulsed Light (IPL) therapy will be performed using the OptiLIGHT® device (Lumenis Be Ltd., Yokneam, Israel). IPL treatment involves the application of high-intensity, non-coherent, polychromatic light within the 500 to 1200 nm wavelength spectrum. Participants will receive 3 IPL sessions over 6 weeks, with sessions targeting the periocular area and upper eyelids to improve meibomian gland function. Each session includes the application of 50 light pulses to the periocular area and upper eyelids using specified parameters (e.g., fluence 14 J/cm² for the periocular area, fluence 11 J/cm² for the upper eyelids).
Drug: Tear Substitute Treatment (Supportive Therapy) — All participants will also receive supportive therapy with tear substitutes throughout the study period. This includes:
  Idroflog® (0.2% Hyaluronic Acid with 0.001% Hydrocortisone): Applied 3 times per day.
  VisuXL gel® (Cross-linked Carboxymethyl Cellulose with Coenzyme Q10): Applied once a day.
  Artelac® Nighttime Gel (0.24% Sodium Hyaluronate with Carbomer): Applied before sleeping. These tear substitutes are intended to provide symptomatic relief and support tear film stability during the treatment period.

SUMMARY:
This study examines the effectiveness of combining Quantum Molecular Resonance (QMR) and Intense Pulsed Light (IPL) treatments for Mixed Dry Eye, a condition where both tear production and tear quality are compromised. Twenty-five patients received both treatments over a period of six weeks, and their symptoms and tear quality were monitored for three months.

DETAILED DESCRIPTION:
Study Title: Efficacy of Quantum Molecular Resonance Combined with Intense Pulsed Light in Mixed Dry Eye: A Prospective Clinical Study

Purpose of the Study: This study aims to evaluate how well two treatments-Quantum Molecular Resonance (QMR) and Intense Pulsed Light (IPL)-work when used together to treat Mixed Dry Eye (MDE). Mixed Dry Eye is a condition that affects both the quantity and quality of tears, leading to discomfort and vision problems. The goal is to see if combining these treatments can better relieve symptoms and improve tear production and stability.

What is Mixed Dry Eye? Dry Eye Disease is a common condition that can cause symptoms like burning, itching, and blurred vision. Mixed Dry Eye occurs when both the tear production is low, and the tears evaporate too quickly, leading to chronic discomfort.

What are QMR and IPL Treatments?

QMR (Quantum Molecular Resonance): This is a newer technology that uses low-intensity, high-frequency waves to stimulate the cells in the eye. It may help improve tear production and reduce inflammation.

IPL (Intense Pulsed Light): This treatment uses light to heat the skin around the eyes, which helps improve the function of glands that produce the oily layer of tears, preventing tears from evaporating too quickly.

Study Design:

Participants: 25 patients with Mixed Dry Eye Treatment: Participants received 4 sessions of QMR and 3 sessions of IPL over 6 weeks. They were also given tear substitutes to use during the study.

Follow-up: Patients were evaluated at the beginning, and after 1 and 3 months to assess the improvement in their condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with Mixed Dry Eye (MDE)
* Ocular Surface Disease Index (OSDI) score of 13 or higher
* Non-Invasive Tear Film Break-Up Time (NIBUT) less than 10 seconds
* Lipid Layer Thickness (LLT) less than 75 nm
* Schirmer I Test (ST) without anesthesia less than 5 mm in 5 minutes

Exclusion Criteria:

* Presence of skin conditions that prevent QMR or IPL treatments
* Corneal disorders that affect diagnostic tests, including:
* Active corneal infections
* Corneal dystrophies
* Active ocular allergy
* Previous device-based dry eye treatments, such as:
* Microblepharoexfoliation
* Low-level light therapy
* Vectored thermal pulsation
* Inability to understand or comprehend the informed consent
* Pregnant or lactating women
* Contact lens wearers who do not discontinue lens use at least one week before baseline and follow-up exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Improvement in Ocular Surface Disease Index (OSDI) Score | Baseline, 1 month, 3 months
  The Ocular Surface Disease Index (OSDI) is a patient-reported questionnaire used to assess the severity of dry eye symptoms. It includes 12 items, with scores ranging from 0 (no symptoms) to 100 (severe symptoms). The change in OSDI score from baseline to 1 month and 3 months after treatment will be measured. A significant reduction in OSDI score indicates an improvement in dry eye symptoms.

SECONDARY OUTCOMES:
Change in Lipid Layer Thickness (LLT) | Baseline, 1 month, 3 months
  Lipid Layer Thickness (LLT) of the tear film will be measured using the Lipiview II ocular surface interferometer. The LLT is expressed in nanometers (nm) and reflects the thickness of the lipid layer in the tear film. The change in LLT from baseline to 1 month and 3 months after treatment will be assessed to determine the effectiveness of the combination therapy in improving tear film stability.
Change in Non-Invasive Tear Film Break-Up Time (NIBUT) | Baseline, 1 month, 3 months
  Non-Invasive Tear Film Break-Up Time (NIBUT) will be measured using the Keratograph 5M. NIBUT is the time taken for the tear film to break up after a blink, without the use of dyes or invasive techniques. It will be recorded in seconds. An increase in NIBUT indicates improved tear film stability. The change in NIBUT will be evaluated from baseline to 1 month and 3 months after treatment.
Change in Schirmer I Test (ST) Score | Baseline, 1 month, 3 months
  The Schirmer I Test (ST) measures tear production. A strip of filter paper is placed under the lower eyelid, and the length of the wet portion of the strip is measured in millimeters after 5 minutes. The test is performed without anesthesia. The change in ST score from baseline to 1 month and 3 months after treatment will be used to assess improvements in tear production.

OTHER OUTCOMES:
Correlation Between Clinical Endpoints and Symptom Improvement | 3 months
  This exploratory outcome measure will analyze the correlation between clinical endpoints (such as NIBUT, LLT, and ST) and the improvement in OSDI scores. The goal is to determine which clinical measures most strongly predict symptom improvement.

CONTACTS AND LOCATIONS:
Overall Officials: José-María Sánchez-González, OD, MsC, PhD, Study Chair — University of Seville; Carlos Rocha-de-Lossada, MD PhD, Study Director — University of Seville
Locations (1):
- Tedesco Eye Center, Girifalco, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality concerns and the lack of a data-sharing agreement in place. However, aggregated results and key findings will be published in peer-reviewed journals.